CLINICAL TRIAL: NCT04045028
Title: A Phase Ia/Ib Open-Label, Multicenter Study Evaluating the Safety and Pharmacokinetics of Tiragolumab as a Single Agent and in Combination With Atezolizumab and/or Daratumumab in Patients With Relapsed or Refractory Multiple Myeloma, and as a Single Agent and in Combination With Rituximab in Patients With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD), and Preliminary Activity of Tiragolumab in Participants With Relapsed or Refractory Multiple Myeloma or With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO41036; 2021-006032-92 (EudraCT Number)
Record Dates: First submitted 2019-07-22; First posted 2019-08-05 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Multiple Myeloma; Non-Hodgkin Lymphoma; B-Cell Lymphoma
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Lymphoma, B-Cell | interventions — Tiragolumab; daratumumab; Rituximab; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A: Tiragolumab R/R MM (Experimental): Participants with relapsed or refractory (R/R) Multiple Myeloma (MM) will receive a single dose of 600 mg tiragolumab by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W).
  Interventions: Drug: Tiragolumab
- Arm B: Tiragolumab R/R NHL (Experimental): Participants with relapsed or refractory (R/R) non-Hodgkin Lymphoma (NHL) will receive a single dose of 600 mg tiragolumab by IV infusion Q3W.
  Interventions: Drug: Tiragolumab
- Arm C: Tiragolumab + Daratumumab R/R MM (Experimental): Participants with R/R MM will receive 600 mg tiragolumab Q3W + daratumumab by subcutaneous (SC) injection.
  Interventions: Drug: Tiragolumab; Drug: Daratumumab/rHuPH20
- Arm D: Tiragolumab + Rituximab R/R NHL (Experimental): Participants with R/R NHL will receive 600 mg tiragolumab Q3W + rituximab by IV infusion and SC injection (optional).
  Interventions: Drug: Tiragolumab; Drug: Rituximab
- Arm E: Tiragolumab + Atezolizumab + Daratumumab R/R MM (Experimental): Participants with R/R MM will receive 600 mg tiragolumab Q3W + atezolizumab by IV infusion Q3W + daratumumab by SC injection.
  Interventions: Drug: Tiragolumab; Drug: Daratumumab/rHuPH20; Drug: Atezolizumab

INTERVENTIONS:
Drug: Tiragolumab — Administered by IV infusion at a fixed dose of 600 mg on Day 1 of each 21-day cycle (Q3W)
Drug: Daratumumab/rHuPH20 — Administered by SC injection 1800 mg/30,000 U rHuPH20 weekly for a total of 6 doses, then every 3 weeks for a total of 16 doses (first dose given at Week 7), then every 4 weeks from Week 55 onward until disease progression
  Arms: Arm C: Tiragolumab + Daratumumab R/R MM; Arm E: Tiragolumab + Atezolizumab + Daratumumab R/R MM
Drug: Rituximab — Administered for a total of 8 doses. Rituximab will be administered by IV infusion for the first dose at a dose of 375 mg/m^2. After administration of at least one full infusion of IV rituximab, the SC formulation of rituximab (rituximab and rHuPH20) may be used for the remaining doses per institutional guidelines. SC rituximab will be administered at a dose of 1400 mg rituximab/23400 U rHuPH20 once weekly (QW).
  Arms: Arm D: Tiragolumab + Rituximab R/R NHL
Drug: Atezolizumab — Administered by IV infusion at a fixed dose of 1200 mg Q3W
  Arms: Arm E: Tiragolumab + Atezolizumab + Daratumumab R/R MM

SUMMARY:
This is a Phase I open-label, multicenter study designed to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary activity of tiragolumab administered as a single agent or in combination with atezolizumab and/or daratumumab or rituximab in participants with relapsed or refractory (R/R) multiple myeloma (MM) or R/R non-Hodgkin lymphoma (NHL).

DETAILED DESCRIPTION:
In the Phase Ia part of the study, tiragolumab is administered as a single agent in participants with R/R MM or R/R NHL.

In the Phase Ib part of the study, tiragolumab is administered in combination with atezolizumab and/or daratumumab in participants with R/R MM or with rituximab in participants with R/R NHL.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria (All Participants):

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of >/= 12 weeks

Inclusion Criteria Specific to Arms A, C and E (R/R MM):

* Arm A only: Must have R/R MM for which no established therapy for MM is appropriate and available or be intolerant to those established therapies
* Arms C and E only: Participants with R/R MM who have received at least 3 prior lines of therapy.
* Measurable disease defined by laboratory test results.

Inclusion Criteria Specific to Arms B and D (R/R NHL):

* Participants with histologically confirmed B-cell NHL who have relapsed or failed to respond to at least two prior systemic treatment regimens and for which no suitable therapy of curative intent or higher priority exists.
* Must have at least one bi-dimensionally measurable lesion.

Exclusion Criteria:

General Exclusion Criteria (All Participants):

* Any anti-cancer therapy, whether investigational or approved, including chemotherapy, monoclonal antibody, radioimmunoconjugate, antibody-drug conjugate, hormonal therapy, and/or radiotherapy, within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to initiation of study treatment
* Prior treatment with any anti-TIGIT agent
* Prior treatment with chimeric antigen receptor-T (CAR-T) therapy within 12 weeks before first study drug administration
* Autologous Stem-Cell Transplantation (ASCT) within 100 days prior to first study drug administration
* Active or history of autoimmune disease or immune deficiency
* Known active bacterial, viral (including SARS-CoV-2), fungal, mycobacterial, parasitic, or other infection at study enrollment, or any major episode of infection within 4 weeks prior to first study drug administration

Exclusion Criteria Specific to Arms A, C and E (R/R MM):

* Primary or secondary plasma cell leukemia
* Current or history of CNS involvement by MM

Exclusion Criteria Specific to Arms B and D (R/R NHL):

* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab
* Current or history of CNS lymphoma
* Current eligibility for ASCT

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events | Through study completion, an average of 1 year
  Determined according to the NCI CTCAE Version 5.0

SECONDARY OUTCOMES:
Serum Concentration of Tiragolumab | Cycles 1, 2, 3, 4, 8, 12, 16, 17 and then every 8 cycles (each cycle is 21 days) and at Treatment Discontinuation Visit (up to 2 years)
Serum Concentration of Atezolizumab | Cycles 1, 2, 3, 4, 8, 12, 16, 17 and then every 8 cycles (each cycle is 21 days) and at Treatment Discontinuation Visit (up to 2 years)
Objective Response Rate (ORR) for R/R MM | Through study completion, an average of 1 year
  Proportion of participants with a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR), as defined by the International Myeloma Working Group (IMWG) criteria
ORR for R/R NHL | Through study completion, an average of 1 year
  Proportion of participants with a CR or PR on two consecutive occasions >/= 4 weeks apart, according to the Lugano classification
Percentage of Participants With Anti-Drug Antibodies (ADAs) to Tiragolumab | Cycles 1, 2, 4, 8, 12, 16, 17 and then every 8 cycles (each cycle is 21 days) and at Treatment Discontinuation Visit (up to 2 years)
Percentage of Participants With ADAs to Atezolizumab | Cycles 1, 2, 4, 8, 12, 16, 17 and then every 8 cycles (each cycle is 21 days) and at Treatment Discontinuation Visit (up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- United States (9):
  - Colorado Blood Cancer Institute (CBCI) at Presbyterian/ St. Luke's Medical Center, Denver, Colorado
  - Emory Clinic, Atlanta, Georgia
  - University of Maryland, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Clinical Research Alliance, Westbury, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - University of Pennsylvania; School of Medicine, Philadelphia, Pennsylvania
  - SCRI, Nashville, Tennessee
  - Virginia Cancer Specialists (Fairfax) - USOR, Fairfax, Virginia
- South Korea (5):
  - Samsung Medical Center; Nephrology Department, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei Cancer Center; Yonsei Uni Coll. Med., Seoul
  - Seoul St.Mary's Hospital; Medical Oncology, Seoul
  - Asan Medical Center; Internal Dept / Gastorenterology, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).